CLINICAL TRIAL: NCT01636050
Title: Phase 1 Study of Child Exercise Training
Brief Title: Effect of Squat Training on Body Composition, Muscular Strength and Motor Fitness for Youth- Randamized Trial
Acronym: CET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Fitness and Sports in Kanoya (Other)
Responsible Party: Principal Investigator, Yohei Takai, assisstant professor, National Institute of Fitness and Sports in Kanoya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CST-002
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Physical Conditioning
Keywords: squat exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Training group (Experimental)
  Interventions: Other: squat exercise training
- Control group (Experimental)
  Interventions: Other: squat exercise training

INTERVENTIONS:
Other: squat exercise training — Intervention may include squat exercise for 8 weeks
  Other Names: school-based exercise training

SUMMARY:
The purpose of this study is to determine the effects of body mass-based squat training on body composition, muscular strength and motor fitness in adolescents.

DETAILED DESCRIPTION:
Body composition Percent body fat by bioimpedance muscle thickness at the thigh anterior by ultrasound

Muscle strength Maximal voluntary knee extension torque by myometer

Motor fitness sprint velocity by non-motorized treadmill Jump height by a matswitch system.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescents

Exclusion Criteria:

* Participants do not have medical and orthopedic disorder.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Percent body fat by bioelectrical impedance | Eight week

SECONDARY OUTCOMES:
knee extension strength by myometer | eight weeks